CLINICAL TRIAL: NCT05949853
Title: Enhanced Respiratory Polygraphy (PV_e) Using Single Channel EEG-based Automatic Sleep Scoring in Suspected Obstructive Sleep Apnea: Feasibility and Efficiency as Compared With Polygraphy and Polysomnography
Brief Title: Enhanced Respiratory Polygraphy in Suspected OSA
Acronym: PVa
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0238
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-07

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Polysomnography; Polygraphy; single channel EEG automated sleep scoring
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients hospitalized at the Center for Sleep and Respiratory Diseases, between 09/2022 and 11/2022 for suspected OSA All these patients underwent a full night polysomnography
  Interventions: Other: the respiratory parameters (AHI) and time spent

INTERVENTIONS:
Other: the respiratory parameters (AHI) and time spent — interpret the recording will be evaluated for PSG, PV and PV+ASEEGA Apnea Hypopnea Index as assessed by PSG (respiratory signals + electro-encephalography + electro-oculography + chin electromyography), PV (respiratory signals) and PV+ASEEGA (respiratory signals + result of sleep stages and arousals scoring by ASEEGA algorithm based on automatic analysis of one EEG Cz-Pz channel)

SUMMARY:
Obstructive Sleep Apnea (OSA) remains underdiagnosed in 2022, as a result of the unawareness of its serious health-related consequences and the lack of diagnosis accessibility. Respiratory polygraphy (PV) is widely used as a screening tool and sometimes a diagnosis test, although polysomnography (PSG) remains the gold standard investigation as it provides complete information about sleep architecture and arousals. Thus, it has been shown that the Apnea Hypopnea Index (AHI) and Respiratory Disorder Index (RDI) are underestimated by PV vs PSG. Approaches to substitute PSG by simpler but equally efficient diagnosis tests have included devices aiming to record complementary signals and to analyze them with Artificial Intelligence. In this context, ASEEGA algorithm has demonstrated its performance for automatic sleep scoring in healthy individuals and patients with various sleep disorders, based on a single channel EEG analysis.

This study aims at comparing the real-life performance and feasibility of added single channel EEG automatic sleep scoring using ASEEGA to PV versus standard PV and PSG in adults referred to a regional sleep reference center for suspected OSA.

We hypothesize that this approach (1) is as accurate as PSG and more accurate that PV for AHI analysis, and (2) is less time-consuming than PSG.

ELIGIBILITY:
Inclusion Criteria:

- Hospitalized at the Center for Sleep Medicine and Respiratory Diseases, Hôpital de la Croix-Rousse, Lyon Academic Hospital, Lyon between 09/2022 and 11/2022 for PSG following suspected OSA .

Exclusion Criteria:

* Unreliable sleep scoring due to artefacts (> 10% of the recording) or to epileptic abnormalities on the electroencephalography recordings
* Presence of other suspected sleep disorder: central hypersomnia, rapid-eye-movement (REM) or non-REM sleep parasomnia, sleep-related motor disorders...
* Ongoing psychotropic medication
* Opposition of the patient to the use of their data.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Hospitalized at the Center for Sleep Medicine and Respiratory Diseases
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Apnea Hypopnea Index as assessed by PSG | analysis will start in January 2023 and should be completed after 6 months.
  Apnea Hypopnea Index will be scored by 2 sleep medical experts at 3 occurrences separated by 1 months interval in a random order (PSG/PV/PV+ASEEGA).
  Apnea Hypopnea Index in the three groups (PSG/PV/PV+ASEEGA) will be compared with Friedmann test or one factor ANOVA for paired data, according to data distribution, for each scorer

CONTACTS AND LOCATIONS:
Locations (1):
- Service de médecine du sommeil et des maladies respiratoires, Lyon, France